CLINICAL TRIAL: NCT00190242
Title: Study of Immunogenicity of Anti-HAV Immunisation in HIV-1 Infected Patients, Co-infected or Not With HBV and/or HCV. HEP.A.VAC Study.
Brief Title: Immunogenicity and Tolerance of Two Strategies of Anti-HAV Vaccination in HIV-infected Patients
Acronym: HEPAVAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ensemble contre le SIDA (Unknown); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P050706
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2005-06

CONDITIONS: HIV Infection
Keywords: HIV; hepatitis A; vaccine; HBV and/or HCV co-infection
MeSH Terms: conditions — HIV Infections; Hepatitis A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group1:3 administrations of Havrix (Experimental): group 1 received immunisation with Havrix (1440IU) at weeks S0, S4, S24
  Interventions: Drug: group1
- group2: 2 administrations of Havrix (Active Comparator): group 2 received usual immunisation with Havrix (1440IU) at weeks S0 and S24
  Interventions: Drug: group2

INTERVENTIONS:
Drug: group1 — Havrix at 1440IU was administrated à weeks S0, S4 and S24
  Arms: group1:3 administrations of Havrix
Drug: group2 — Havrix (1440IU) was administrated at weeks S0 and S24 according to RECOMMANDATIONS
  Arms: group2: 2 administrations of Havrix

SUMMARY:
Immunogenicity is reduced in immunocompromised patients. The aim of this prospective randomized study is to evaluate tolerance and immunogenicity of 2 doses versus 3 doses of anti-HAV vaccine in HIV-1 infected patients with CD4 count between 200 and 500 per mm3, co-infected or not with HBV and/or HCV. The factors influencing vaccine immunogenicity will be evaluate.

DETAILED DESCRIPTION:
RECOMMANDATIONS for hepatitis A vaccination is the same for HIV-infected patients than for general population. However, immunogenicity induced with 2 doses of anti-HAV vaccine is lower in HIV-infected patients. The primary objective of the study is to compare the immunogenicity (percentage of patients with anti-HAV antibodies > 20 mUI/ml at month 7) of 2 strategies (2 doses at months 1 and 6, versus 3 doses at months 1, 2 and 6)of anti-HAV vaccine in HIV-1 infected patients co-infected with HBV and/or HCV with CD4 cell count between 200 and 500/mm3. The second objectives are to compare mean anti-HAV antibodies titers obtained with the 2 strategies, the durability of the seroprotection 12 months after the end of vaccination, and the safety. The PARAMATERS than may have an effect on the immune response will be evaluated.

This open, prospective, study have included 99 patients, aged from 18 to 55 years old. Patients were randomized to receive 2 or 3 doses of HAVRIX 1440 UI intramuscularly at week O, 4, and 24 or week 0, and 24. Clinical and biological safety is evaluated after each immunisation and blood samples for serological evaluation taken at week -4, 4, 8, 24 and 28 for immunogenicity and week 72 for long term analysis

ELIGIBILITY:
Inclusion Criteria:

* VIH-1 infection, aged 18-55 years negative anti-HAV IgG CD4 cell count between 200 and 500/mm3

Exclusion Criteria:

* prior anti-HAV vaccination immunosuppressive treatment splenectomy Prothrombin time < 50%, platelets< 50 000/mm3 fever serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) activity > 2 ULN for non co-infected patients, > 5 ULN for co-infected patients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2003-06; Primary Completion 2006-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
percentage of patients with anti-HAV antibodies superior 20 mUI/ml 7 months after the first vaccination | during de study
  percentage of patients with anti-HAV antibodies superior 20 mUI/ml 7 months after the first vaccination

SECONDARY OUTCOMES:
anti-HAV antibodies mean geometric titers 7 months after the first vaccination | during the study
  anti-HAV antibodies mean geometric titers 7 months after the first vaccination
durability of seroprotection 1 year after the end of vaccination | during the study
  durability of seroprotection 1 year after the end of vaccination
safety | during the study
  safety
predictive factors of vaccinal response | during the study
  predictive factors of vaccinal response

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Sophie GRABAR, MD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - CIC de vaccinologie Cochin Pasteur, Service de médecine interne, hôpital Cochin, Paris
  - CISIH, Hôpital de Strasbourg, Strasbourg